CLINICAL TRIAL: NCT05696496
Title: Évaluation d'un Dispositif de détection du Sommeil " Easy Sleep Monitoring " (ou " Couette Intelligente ") Par Rapport à la vidéo-polysomnographie, Chez Des Patients Avec Des Troubles du Sommeil et Des Sujets Sains
Brief Title: Evaluation of e New Sleep Detection Device "Easy Sleep Monitoring"
Acronym: ESM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2022 FANTINI
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Sleep Disorder
Keywords: video polysomnography; new sleep detection device
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: the 2 groups (patients with Sleep Disorder Group (TS+) and the control group (TS-)) will receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with sleep disorders (TS+) (Experimental): video polysomnography; the new ESM "intelligent duvet" device
  Interventions: Device: night recording
- control group without sleep disorder (TS-) (Experimental): video polysomnography; the new ESM "intelligent duvet" device
  Interventions: Device: night recording

INTERVENTIONS:
Device: night recording — The patients/controls will arrive in the evening at the Sleep Laboratory (Functional Exploration Department of the Nervous System of the Clermont-Ferrand University Hospital) to carry out complete vPSG and test the new ESM "intelligent duvet"device. A qualified technician will place the electrodes according to the procedures usually followed at the Sleep Center for vPSG recording. The ESM duvet will be placed on the patient's body as a blanket, instead of the blankets normally provided by the hospital. Patients/controls will be monitored overnight by an infrared video camera.

SUMMARY:
If the video-polysomnographic (vPSG) recording in the laboratory remains the reference examination in Sleep Medicine Centers for the diagnosis of sleep pathologies, the high prevalence of sleep disorders in the general population and the growing demand for exploration and management may require the use of alternative techniques such as new sleep recording or analysis devices. In collaboration with the Creative Mechatronics Company (Issoire) and the Ennery Confection Company (Le Puy en Velay), we have developed a "portable" sleep detection prototype called Easy Sleep Monitoring (ESM) which consists of an "intelligent" duvet equipped with a series of sensors capable of detecting movements and, through this, estimating sleep duration and quantifying motor phenomena during sleep. Indeed, it is a duvet which has in its thickness a grid of 35 electronic cards, equipped with an actimetric sensor and a temperature sensor. The distribution of the sensors makes it possible to detect the motor activity of the sleeper on all the body regions by considerably increasing the sensitivity and specificity compared to actimetry at the wrist.

The advantage of this duvet compared to other "wearable" devices is represented by its ease of use, being less restrictive, having a reduced implementation time and not requiring the user's collaboration. For example, it could be used for sleep monitoring in the elderly and/or in a situation of hypomobility in the context of Residential establishment for dependent elderly people or hospitals. At home, it could be a sleep monitoring tool, such as monitoring treatment for insomnia, medicinal or not, or to monitor motor activity during sleep, as in the monitoring of nocturnal akinesia in parkinsonian patients.

The main objective of this study is to evaluate the concordance of sleep data obtained with the ESM duvet with those obtained by video-polysomnography (vPSG). Indeed, the vPSG is the gold standard examination in the study of sleep, the only one capable of exactly defining the different stages of sleep and precisely quantifying sleep disorders.

DETAILED DESCRIPTION:
Type of study : monocentric study, a proof of concept study of a new device for sleep detection "Easy Sleep Monitoring" (ESM). This is a category 4.4 clinical investigation with a non-CE marked medical device used in its indication, without the objective of CE marking or establishing compliance

Number of centers: 1

Patients:

This study will be perdormed in 50 subjects (25 patients with sleep disorders (TS+) + 25 subjects without proven sleep disorders (TS-))

Study performance:

Each subject will have 2 visits:

1. First visit (baseline, inclusion visit, 30 minutes) which will include:

   * Information and collection of written consent
   * Recording of demographic and clinical data (age, sex, duration of disease progression, current treatments, medical and surgical history)
   * Pittsburgh PSQI Sleep Quality Index (for TS- group only)
   * Verification of inclusion and non-inclusion criteria.
2. Visit 2 (Month 6) (duration 1 night): The patients/controls will arrive in the evening at the Sleep Laboratory (Functional Exploration Department of the Nervous System of the Clermont-Ferrand University Hospital) to carry out complete vPSG and test the new ESM "intelligent duvet" device.

ELIGIBILITY:
Inclusion Criteria:

For Sleep Disorder Group (TS+):

* Men or women, aged 18 to 85
* With a suspected sleep disorder (sleep apnea, restless legs syndrome RLS, syndrome of periodic leg movements during MPJS sleep, REM sleep behavior disorder, Parkinson's disease, Narcolepsy, etc.), requiring a confirmation of the diagnosis in vPSG.
* Cooperation and understanding to strictly comply with the conditions set out in the protocol - Acceptance of the protocol and signing of a written consent
* Affiliation to the social security system

For Control Group (TS- ):

* Men or women, aged 18 to 85
* Having no sleep disorder: the Pittsburgh PSQI sleep quality index (Buysse et al., 1989) must be <5.
* Cooperation and understanding to strictly comply with the conditions set out in the protocol - Acceptance of the protocol and signing of a written consent
* Affiliation to the social security system

Exclusion Criteria:

For Group TS+ and TS-:

* Patients under guardianship or curatorship or safeguard of justice
* Pregnant or breastfeeding women (given the low risk incurred, the verification will be done on simple declaration of the patient)
* Patients with active implants
* during a period of exclusion from another study,
* refusing to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Effective sleep duration (in minutes) | Month 6
  evaluated by vPSG
Effective sleep duration (in minutes) | Month 6
  evaluated by ESM device

SECONDARY OUTCOMES:
Time spent in bed (in minutes) | Month 6
  evaluated by vPSG
Time spent in bed (in minutes) | Month 6
  evaluated by ESM device
Sleep efficiency (Total sleep time/Time spent in bed) | Month 6
  evaluated by vPSG
Sleep efficiency (Total sleep time/Time spent in bed) | Month 6
  evaluated by ESM device
Sleep latency (in minutes) | Month 6
  evaluated by vPSG
Sleep latency (in minutes) | Month 6
  evaluated by ESM device
Duration of sleep stages (Deep Wave Sleep vs. Paradoxical Sleep)(in minutes) | Month 6
  evaluated by vPSG
Duration of sleep stages (Deep Wave Sleep vs. Paradoxical Sleep) (in minutes) | Month 6
  evaluated by ESM device
% of sleep stages (Deep Wave Sleep vs. Paradoxical Sleep) | Month 6
  evaluated by vPSG
% of sleep stages (Deep Wave Sleep vs. Paradoxical Sleep) | Month 6
  evaluated by ESM device
Number of alarm clocks | Month 6
  evaluated by vPSG
Number of alarm clocks | Month 6
  evaluated by ESM device
Number of position changes | Month 6
  evaluated by vPSG
Number of position changes | Month 6
  evaluated by ESM device
Duration of periodic movements of the lower limbs (in minutes) | Month 6
  evaluated by vPSG
Duration of periodic movements of the lower limbs (in minutes) | Month 6
  evaluated by ESM device
Duration of Cheyne-Stokes periodic breathing (in minutes) | Month 6
  evaluated by vPSG
Duration of Cheyne-Stokes periodic breathing (in minutes) | Month 6
  evaluated by ESM device
number of obstructive and central apneas | Month 6
  evaluated by vPSG
number of obstructive and central apneas | Month 6
  evaluated by ESM device

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, UMR INSERM 1107, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No